CLINICAL TRIAL: NCT00455715
Title: A Placebo-Controlled Single-Dose Trial of Sildenafil in Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Donald Goff, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2005-P-000529
Record Dates: First submitted 2007-04-02; First posted 2007-04-04 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Cognition; Sildenafil; PDE5 Inhibitor
MeSH Terms: conditions — Schizophrenia | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sildenafil — 1 capsule Sildenafil 50mg or Sildenafil 100mg or placebo taken at the time of study visit.
  Other Names: Viagra

SUMMARY:
The study is a double-blind, placebo-controlled, random-order, single-dose crossover trial of sildenafil 50 & 100 mg added to stable antipsychotic treatment in schizophrenia patients to assess whether this PDE5 inhibitor improves cognitive functioning (including verbal memory, fluency, attention, spatial memory, motor speed, and executive function) and clinical symptoms (psychotic, negative, mood symptoms, and self-reports of side-effects).

DETAILED DESCRIPTION:
Specific Aims:

1. Evaluate the effects of single doses of sildenafil 50 & 100 mg compared to placebo on cognitive functioning, including verbal memory, fluency, attention, spatial memory, motor speed, and executive function.
2. Evaluate the effects of single doses of sildenafil 50 & 100 mg compared to placebo on psychotic, negative, and mood symptoms.
3. Assess self-reports of side effects of sildenafil 50 & 100 mg.

Location and Subjects:

25 adult outpatients with schizophrenia will be recruited from the Massachusetts General Hospital outpatient clinic or the Freedom Trail Clinic of the Lindemann Center. All research procedures will be performed at the Psychopharmacology Clinic of the Massachusetts General Hospital. Subjects must be English speaking because the cognitive battery has only been validated in English.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of schizophrenia, any subtype.
2. Age 18-65 years
3. Male or female
4. Clinically stable without a medication change within 4 weeks
5. Able to complete cognitive testing (must be English-speaking)
6. Willing to use appropriate birth control during study participation (if female)

Exclusion Criteria:

1. Active substance abuse or dependence
2. PDE 5 inhibitor taken within 24 hours of study drug
3. Currently taking a drug that inhibits hepatic cytochrome P450 3A4 (eg. Nefazadone, fluvoxamine, erythromycin, ketoconazole, itraconazole, cimetidine, saquinavir, ritonavir, St. John's wort, or grapefruit juice).
4. Currently taking drugs that induce P45 3A4 (eg. phenytoin, carbamezapine, Phenobarbital, rifampin)
5. Unstable medical disease
6. Significant cardiac disease
7. Bleeding disorder
8. Peptic ulcer disease
9. Hepatic impairment
10. Moderate or greater renal impairment
11. History of migraines
12. Currently taking nitrates or alpha blockers
13. Resting blood pressure < 90/50 or >140/90 mm.
14. History of intolerance to PDE5 inhibitors
15. History of inappropriate sexual behavior (eg, masturbation in public, stalking, assault)
16. History of priapism
17. Pregnant or lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-02; Primary Completion 2007-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Evaluate the effects of single doses of sildenafil 50 & 100 mg compared to placebo on cognitive functioning, including verbal memory, fluency, attention, spatial memory, motor speed, and executive function. | 12 days

SECONDARY OUTCOMES:
Evaluate the effects of single doses of sildenafil 50 & 100 mg compared to placebo on psychotic, negative, and mood symptoms. | 12 days
Side effects of sildenafil 50 & 100 mg as self-reported by subjects and as measured with vital signs. | 12 days

CONTACTS AND LOCATIONS:
Overall Officials: Donald C Goff, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Goff DC, Cather C, Freudenreich O, Henderson DC, Evins AE, Culhane MA, Walsh JP. A placebo-controlled study of sildenafil effects on cognition in schizophrenia. Psychopharmacology (Berl). 2009 Jan;202(1-3):411-7. doi: 10.1007/s00213-008-1278-5. Epub 2008 Aug 21. PMID 18716761